CLINICAL TRIAL: NCT06788080
Title: Optimization of Biotinylation Protocol for Next Generation Studies of Red Blood Cell Survival and Function After Transfusion
Brief Title: Optimization of Biotinylation Protocol for Studies of Red Blood Cell Survival and Function After Transfusion
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Vitalant Research Institute (Other)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 11735-01
Record Dates: First submitted 2023-06-16; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Measuring Red Blood Cell Survival After Transfusion
Keywords: Biotin; Red blood cell; Transfusion

STUDY DESIGN:
Intervention Model Description: Each participant will receive BioRBCs labeled with two different doses of biotin and stored for 6h and 24h.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- BioRBC arm (Experimental): Each subject will receive biotin labeled red blood cells stored for 6 hours and 24 hours (two separate aliquots infused sequentially).
  Interventions: Drug: BioRBC

INTERVENTIONS:
Drug: BioRBC — Autologous biotin-labeled RBCs will be transfused to study participants

SUMMARY:
The goal of this clinical trial is to compare two methods of labeling red blood cells with biotin. The main question to answer is whether red blood cells labeled 48 hours before transfusion survive as long as red blood cells labeled 6 hours before transfusion. Secondary questions are to measure the quality of the red blood cells and whether or not the biotin-labeled red blood cells induce antibodies in transfusion recipients.

This study participant will have six study visits:

1. Screening visit, collect 35 ml blood, about 3 tablespoons
2. Donate 500 ml blood
3. Receive 20 ml of biotin labeled blood transfusion, collect 40 ml blood, about 3 tablespoons
4. Return 1 day after transfusion for blood draw (25 ml, about 2 tablespoons)
5. Return 30 days after transfusion for blood draw (25 ml, about 2 tablespoons)
6. Return 90 days after transfusion for blood draw (25 ml, about 2 tablespoons)

DETAILED DESCRIPTION:
The objective of this open label, pilot, single center, trial of biotinylated red blood cells (BioRBCs) is to determine the impact of RBC biotinylation timing (48h vs 6h prior to transfusion) on autologous BioRBCs posttransfusion recovery in 12 healthy subjects. The rationale is to determine the feasibility of manufacturing BioRBC at a central site that is remote from the site of the clinical study, where transfusion occurs. Manufacturing and transportation will result in a delayed (up to 48 hrs.) transfusion of the BioRBCs. In this trial each subject will donate one unit of autologous whole blood which will be manufactured into leukoreduced packed RBCs (pRBCs) in additive solution-1 (AS-1) and stored for 42 days. Biotin labelling of the pRBCs will occur at 2 different time points, after 35-40 days of storage or after 37-42 days of storage with 2 different doses of biotin (3 µg/mL vs 15 µg/mL). Subjects will be stratified at the time of enrollment (first 6 subjects enrolled vs last 6 subjects enrolled) to a labelling sequence related to both the dose of biotin label and the time of labelling. The stratification sequence is defined by subjects with an earlier enrollment (first 6 subjects enrolled) who will have low dose biotin label (3µg/mL) after storage of autologous pRBCs at the earlier time point (35-40 days), and the high dose biotin label (15µg/mL) after storage of autologous pRBCs at the later time point (37-42 days). The alternative labelling procedure, for subjects enrolled later on study (last 6 subjects enrolled), will utilize the high dose biotin label (15 µg/mL) after storage of autologous pRBCs at the earlier time point (35-40 days) and the low dose biotin label (3µg/mL) after storage of autologous pRBCs at the later time point (37-42 days).

This stratification is designed to result in the second biotin labelling to occur on the day of transfusion (which is also approximately 2 days after the first biotinylation process). Thus, each subject will receive a total of two sequential 10 mL doses of BioRBCs during one infusion visit.

ELIGIBILITY:
Inclusion Criteria:

Age 18 years or older;

Self-report that he or she feels well and healthy;

Be able and willing to provide written informed consent;

Be available for the duration of the trial (up to 28 weeks) and able to come to the treatment clinic for scheduled trial visits. This includes screening up to a month before blood donation, a blood donation, BioRBC transfusion (37-42 days after blood donation), and follow up visits 24h, 30 and 90 days after transfusion.

Females should either be surgically sterile (hysterectomy or tubal ligation) or should use a highly effective, medically accepted contraceptive regimen. Highly effective methods of birth control are defined as those that result in a lower failure rate (i.e., less than 1% per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, intrauterine devices, sexual abstinence, condoms with spermicide, or vasectomized partner.

All females must have a negative pregnancy test prior to enrollment. Post-menopausal females (women over 50 years of age who, in the absence of pregnancy, have a minimum of 2 months without menses) and females who have had a hysterectomy or oophorectomy will not be tested; and

Understand the English language.

Exclusion Criteria:

Other previously diagnosed RBC disorders (sickle cell disease, thalassemia, spherocytosis, hemoglobin variants);

Other severe acute or chronic medical or laboratory abnormality that may increase the risk associated with study participation or investigational process administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the individual inappropriate for entry into this study or would prevent completion of the study;

Participation in another research study with an investigational drug within four weeks prior to or during the planned study duration;

Positive screen for anti-BioRBC antibodies detectable using ID-MTS Gel Cards (Ortho Clinical Diagnostics);

Known liver, kidney, cardiovascular, neurologic, gastrointestinal, blood, endocrine/metabolic, autoimmune or pulmonary disease, or untreated hypertension;

Cancer of any kind (except basal cell) under treatment;

Known or past coagulopathy conditions;

Any medical conditions or medications on the AABB medical deferral list;

Known HIV or acquired immunodeficiency syndrome-related illness or received a positive test result for HIV infection;

Positive test for hepatitis B virus, hepatitis C virus, human T-cell lymphotropic virus (HTLV), West Nile virus, or syphilis;

History of significant treated or untreated mental health issues;

Female subject who is pregnant, lactating, or with a positive pregnancy test;

Currently taking an antibiotic or another medication for an infection;

Known intolerance to any components (biotin) in the investigational drug formulation;

Systolic blood pressure > 140 mm Hg;

Diastolic blood pressure > 90 mm Hg;

Temperature > 100°F;

Known hemoglobin <13 for male donors and <12.5 for female donors;

Positive direct antiglobulin test (DAT);

Treatment with any investigational agent within 1 month before treatment infusion for this trial;

Unwilling or unable to comply with the requirements of this protocol, including the presence of any condition (physical, mental, or social) that is likely to affect the subject's return for follow-up visits on schedule;

Other unspecified reasons that, in the opinion of the investigator, make the subject unsuitable for enrollment;

Institutionalized because of legal or regulatory order

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-03-07 (Actual); Primary Completion 2024-11-04 (Actual); Study Completion 2024-11-04 (Actual)

PRIMARY OUTCOMES:
Percent BioRBC recovery | 24 hours after transfusion
  The percent recovery of BioRBCs (the percentage of infused BioRBCs remaining in circulation) labeled 48 hours vs. 6 hours prior to transfusion will be tested in each participant. Recovery will be compared between BioRBCs labeled at 6 vs. 48 hours.

SECONDARY OUTCOMES:
Percent BioRBC recovery | 10 min, 30 min, 1 hour, 30 days, and 90 days after transfusion
  The percentage recovery of BioRBCs (the percentage of infused BioRBCs remaining in circulation) labeled 48 hours vs. 6 hours prior to transfusion will be tested in each participant. Recovery will be compared between BioRBCs labeled at 6 vs. 48 hours.
Number of participants who form BioRBC antibodies | Pre-transfusion and 1, 30, and 90 days after transfusion
  Test for the presence of antibodies directed against BioRBCs using a gel card assay. Results will be positive or negative, and we will track the number of participants with positive results.
Percent of cells with BioRBC oxidative stress | 10 min, 30 min, 1 hour, 1 day, 30 days, and 90 days after transfusion
  Measure BioRBC oxidative stress by staining cells with BODIPY. Results will be expressed as the percentage of BODIPY+ BioRBCs in each participant. BODIYP+ BioRBCs will be compared between BioRBCs labeled at 6 vs. 48 hours.
Percent of BioRBCs expressing phosphatidyl serine | 10 min, 30 min, 1 hour, 1 day, 30 days, and 90 days after transfusion
  Measure BioRBC phosphatidyl serine expression, which will be measured as the percentage of BioRBCs that bindannexin V, assessed by flow cytometry. Annexin V+ BioRBCs will be compared between BioRBCs labeled at 6 vs. 48 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Norris, MD, Principal Investigator — Vitalant Research Institute
Locations (2):
- United States (2):
  - Anschutz Medical Center, Aurora, Colorado
  - Vitalant Research Institute, Denver, Colorado

IPD SHARING:
Plan to Share IPD: Yes
A de-identified study dataset will be submitted to Westat, the Data Coordinating Center (DCC) for the REDS-IV-P program. Study outcomes (post-transfusion RBC recovery, BioRBC antibody status, and annexin V and RBC redox state will be outcomes reported). The DCC will create public use datasets and deliver them to NHLBI at the end of the study (and end of the REDS-IV-P program).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: At the end of the REDS-IV-P program, estimated in March 2026, the public use data sets will be available and will be available. The DCC will maintain a data archive for three years following the end of the REDS-IV-P contract (through March 21, 2029). At that point, data not on the NIH website will be destroyed.
Access Criteria: Investigators can email the principal investigator to obtain access to the data and study protocol.

REFERENCES:
- [Background] Donnenberg AD, Kim-Shapiro DB, Kanias T, Moore LR, Kiss JE, Lee JS, Xiong Z, Wang L, Triulzi DJ, Gladwin MT. Optimizing interpretation of survival studies of fresh and aged transfused biotin-labeled RBCs. Transfusion. 2023 Jan;63(1):35-46. doi: 10.1111/trf.17192. Epub 2022 Dec 9. PMID 36494878
- [Background] Mock DM, Stowell SR, Franco RS, Kyosseva SV, Nalbant D, Schmidt RL, Cress GA, Strauss RG, Cancelas JA, von Goetz M, North AK, Widness JA. Antibodies against biotin-labeled red blood cells can shorten posttransfusion survival. Transfusion. 2022 Apr;62(4):770-782. doi: 10.1111/trf.16849. Epub 2022 Mar 11. PMID 35274303